CLINICAL TRIAL: NCT00233584
Title: A Study to Evaluate the Feasibility of a Treatment Algorithm in Newly Diagnosed Asthmatic Children. An Open Follow-up to Asthma Prevention in Infants/Young Children (PAC)
Brief Title: Pulmicort Asthma Prevention (Post-PAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5254C00004
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Asthma
Keywords: Children of asthmatic mothers
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Procedure: Pulmicort (budesonide) pMDI

SUMMARY:
This prospective study will evaluate the feasibility of the defined decision tree for the treatment of asthmatic young children. Children who develop episode (=3 consecutive days) of any troublesome lower respiratory symptoms are treated according to a strictly pre-defined multi-steps treatment algorithm until the age of 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Children form the COPSAC/PAC study with episodes of troublesome respiratory symptoms. Episodes are defined as 3 consecutive days of any troublesome lower respiratory symptoms.

Exclusion Criteria:

* Differential diagnoses including at least a chest x-ray and sweat test.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 2001-07; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Success rate of the treatment algorithm: Frequency of protocol deviations, asthma exacerbations, different treatment steps.
Efficacy - development of lung function.

SECONDARY OUTCOMES:
Acceptability of the treatment algorithm by the parents.
Growth rate and BMD.
Exhaled nitrogen Oxide, bronchohyperresponsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Denmark Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Copenhagen, Denmark